CLINICAL TRIAL: NCT05478330
Title: Evaluation of Efficacy of Topical Flutamide in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Essam, Lecturer of Dermatology, Zagazig University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 6597
Record Dates: First submitted 2022-07-14; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Acne Vulgaris Superficial Mixed Comedonal and Inflammatory
MeSH Terms: interventions — Flutamide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Flutamide group) (Experimental): Flutamide was supplied in the form of yellow powder and obtained from Sigma Pharmaceutical Industries, Egypt.
  Tween 80 and Propylene glycol were obtained from Sigma Pharmaceutical Industries, Egypt.
  Oleic acid was purchased from El Gomhouria Company for Trading Chemicals and Medical Appliances, Egypt.
  Interventions: Drug: Flutamide 1% gel
- Group B (control group) (Placebo Comparator): Tween 80 and Propylene glycol were obtained from Sigma Pharmaceutical Industries, Egypt.
  Oleic acid was purchased from El Gomhouria Company for Trading Chemicals and Medical Appliances, Egypt.
  Interventions: Drug: topical gel without flutamide

INTERVENTIONS:
Drug: Flutamide 1% gel — Group A: Flutamide-treated patients: Consisted of 25 patients with acne vulgaris treated with 1% Flutamide topical gel on the face two times per day for a duration of 8 weeks.
  Arms: Group A (Flutamide group)
Drug: topical gel without flutamide — Group B: Consisted of 25 patients with acne vulgaris treated with topical gel with the same component as the other group, except for flutamide, on the face twice per day for a duration of 8 weeks.
  Arms: Group B (control group)

SUMMARY:
From the obtained results, topical Flutamide 1% gel can be a promising, effective, and safe alternative in treating patients with acne vulgaris with minimal side effects.

DETAILED DESCRIPTION:
Flutamide is a non-steroidal anti-androgen, which is used to treat patients with prostate cancer. Due to its anti-androgenic properties can be used in cases of acne, hirsutism, and androgenic alopecia with successful outcomes. To minimize the unnecessary systemic side effects associated with the oral administration of Flutamide. It has been shown that the topical delivery of Flutamide can allow high drug levels at the site of action, decreasing the systemic side effects and improving patient compliance.

The Flutamide group received topical Flutamide 1% gel twice daily on the face for 8 weeks and the control group received the same gel components, without flutamide, twice daily on the face for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Fifty adult patients with acne having inflammatory (papules and pustules) and non-inflammatory (comedones) of different sizes, distribution, and durations were included in this study.

Exclusion Criteria:

* Patients with a history of acne treatment with systemic or topical antibiotics, retinoids, or hormonal therapy within the last 3 months.
* Patients with a history of chronic renal failure, hepatic insufficiency

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
changes in the number of comedones, papules, and pustules | up to 8 weeks
  Response to treatment was evaluated by the changes in the number of comedones, papules, and pustules and by a photographic comparison taken at Baseline ( before treatment) and at 2,4,6, and 8 weeks at (termination of therapy).

SECONDARY OUTCOMES:
side effects | 8 weeks
  scaling, stinging, erythema, dryness

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Essam, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: No